CLINICAL TRIAL: NCT01825954
Title: A Double-Blinded, Randomized, Sham-Controlled, Proof of Concept Study Exploring the Safety and Efficacy of RINCE Technology for the Treatment of Patients With Fibromyalgia
Brief Title: Prospective Evaluation of RINCE to Reduce Fibromyalgia Effects - St. Joseph Mercy Oakland
Acronym: PERRFECT-SJMO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cerephex Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NPT-201
Record Dates: First submitted 2013-04-01; First posted 2013-04-08 (Estimated); Last update posted 2015-09-17 (Estimated); Status verified 2015-09

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Pain; Brain; Stimulation; Device
MeSH Terms: conditions — Fibromyalgia; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- 12-week RINCE (Active Comparator): RINCE - active RINCE therapy involving 24 total treatment applications from NeuroPoint device
  Interventions: Device: RINCE
- 8-week RINCE (Active Comparator): RINCE - active RINCE therapy involving 16 total treatment applications from NeuroPoint device, followed by 8 sham applications from the NeuroPoint device
  Interventions: Device: RINCE
- Sham RINCE (Sham Comparator): Sham RINCE - sham RINCE therapy involving 24 total sham applications from NeuroPoint device
  Interventions: Device: RINCE

INTERVENTIONS:
Device: RINCE — The intervention uses the NeuroPoint device to deliver repeat applications of RINCE therapy stimulation. The sham uses the NeuroPoint device, but the RINCE therapy stimulation is not turned on.
  Other Names: RINCE therapy; RINCE therapy delivered by the NeuroPoint device

SUMMARY:
The purpose of this study is to test the safety and efficacy of a noninvasive cortical electrostimulation therapy known as "Reduced Impedance Noninvasive Cortical Electrostimulation" (RINCE) in the management of fibromyalgia. Patients who meet the 1990 American College of Rheumatology criteria for fibromyalgia will receive up to 24 RINCE treatments delivered by a medical device called "NeuroPoint". Approximately 45 fibromyalgia patients will be randomized into one of three study groups. One of these groups will receive sham treatment, meaning they will receive no treatment at all, while the remaining two groups will receive different amounts of RINCE therapy. The study's primary outcome measure will be the patient's change from baseline in self-reported 24-hour average pain intensity. The study's hypothesis is that there will be a difference between treatment groups in primary outcome measure.

ELIGIBILITY:
Inclusion Criteria:

* Patient must provide written informed consent and privacy authorization prior to participation in the study. Patient must have the ability to read and/or follow written and oral instructions, abide by the study restrictions, and agree to return for the required assessments.
* Patient is male or female, 22-65 years of age (inclusive) at the time of consent.
* Patient must have a confirmed diagnosis of fibromyalgia meeting the ACR 1990 classification criteria for fibromyalgia.
* Patients must have a 24-hour recall pain intensity score at both the screening and baseline visits between 40 and 90 inclusive on a 100 mm VAS scale.
* Female patients of childbearing potential must be willing to use an acceptable method of birth control for the duration of their study participation. Acceptable birth control includes a vasectomized partner, contraceptives (oral, parenteral, or transdermal), intrauterine device, or double barrier method including condoms, sponge, diaphragm, or vaginal ring with spermicidal jellies or cream. Patients considered not of childbearing potential must be surgically sterile (total hysterectomy, bilateral salpingo-oophorectomy, or tubal ligation) or greater than one year post-menopausal, defined as a complete cessation of menstruation for at least one year.
* Patients must be willing to refrain from all excluded therapies for the duration of the study.
* In the opinion of the Investigator, the patient is willing and able to comply with all protocol-specified requirements.

Exclusion Criteria:

* Patient has a current significant psychological or psychiatric disorder (e.g., severe, unstable or poorly controlled depression, severe anxiety or obsessive-compulsive disorder; history of suicide attempt within preceding 5 years or suicidal ideation within preceding 6 months; or any history of bipolar disorder, schizophrenia, schizoaffective or other psychotic disorder).
* Patient has a score of 2 or 3 on item 9 of the BDI, or, based on the investigator's judgment, the patient is at risk of suicidal ideation or behavior.
* Patient is currently using prohibited medications or treatments (see Prohibited Concomitant Therapy section of protocol) including FDA-approved fibromyalgia treatments, other centrally active analgesics, stimulants, anesthetic patches, CPAP and/or TENS therapy.
* Patient has an active diagnosis and is being treated for chronic infection or chronic condition such as lupus, rheumatoid arthritis, Parkinson's disease, multiple sclerosis, hepatitis, polio, seizures, or cancer (other than basal or squamous cell skin cancer).
* Patient has any other chronic pain condition other than fibromyalgia that, in the Investigator's opinion, would interfere with the assessment of fibromyalgia (e.g., rheumatoid arthritis, post herpetic neuralgia, pain associated with diabetic neuropathy, severe pain due to degenerative joint disease, etc.)
* Patient has history of seizure disorder, dementia or epilepsy anytime during his or her life except pediatric febrile seizures.
* Female patient who is pregnant, planning a pregnancy, or breastfeeding.
* Patient has any other disease or medical condition that, in the opinion of the investigator, would interfere with the evaluation of study device efficacy or safety, or would compromise the patient's ability to participate in or complete the study.
* Patient has a history of other cranial electrical stimulation device use, or electroconvulsive therapy.
* Patient has any metal implant, such as stents, aneurysm clips, shunts, pacemakers, defibrillators or neurostimulators. Long-bone implants are not excluded.
* Any anticipated need for surgery that might confound results or interfere with patient's ability to comply with the protocol.
* Myocardial infarction during preceding 12 months, uncontrolled hypertension, active cardiac disease (American Heart Association Functional Class 2, 3 or 4 or Objective Class C or D), clinically significant cardiac rhythm or conduction abnormality, or anticipation of bypass or other cardiac surgery within the next 12 months.
* Current systemic infection (e.g., HIV, hepatitis).
* Patients receiving systemic corticosteroids (> 5 mg prednisone or equivalent per day).
* Patients receiving regular or frequent opioids, opiates or narcotics.
* Pending or current litigation or disability claim (including Workman's Compensation). Patients currently receiving disability benefits will require medical monitor approval on a case-by-case basis.
* Patient has history of alcohol and/or drug abuse.
* Patient has participated in any investigational study within 30 days prior to Screening visit or is currently participating in another clinical trial.
* Patient has received any prior experimental treatment or therapy that, in the opinion of the medical monitor, would compromise the patient's ability to participate in the study.
* Patient is a staff member or relative of a staff member at either the investigative site or the Cerephex Corporation.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2013-03; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in patient 24-hour recall average pain intensity | Assessed at 12 weeks
  Pain intensity evaluated on a 100-mm visual analog scale (VAS)

SECONDARY OUTCOMES:
Patient self-reported Global Impression of Change | Assessed at 12 weeks
Change from baseline in Revised Fibromyalgia Impact Questionnaire | Assessed at 12 weeks
Change from baseline in patient 7-day recall average pain intensity | Assessed at 12 weeks
  Pain intensity evaluated on a 100-mm visual analog scale (VAS)
Change from baseline in Jenkins Sleep Questionnaire | Assessed at 12 weeks
  Sleep measures evaluated using a 100-mm visual analog scale (VAS)

OTHER OUTCOMES:
Change from baseline in Beck Depression Inventory (BDI-II) | Assessed at 12 weeks
Change from baseline in EEG measures | Assessed at 12 weeks
  Various measures collected from resting electroencephalogram (EEG)
Change from baseline in Multiple Ability Self-Report Questionnaire (MASQ) | Assessed at 12 weeks
Change from baseline in Mental Clutter Scale (MCS) | Assessed at 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- St. Joseph Mercy Oakland, Pontiac, Michigan, United States

REFERENCES:
- [Background] Hargrove JB, Bennett RM, Simons DG, Smith SJ, Nagpal S, Deering DE. A randomized placebo-controlled study of noninvasive cortical electrostimulation in the treatment of fibromyalgia patients. Pain Med. 2012 Jan;13(1):115-24. doi: 10.1111/j.1526-4637.2011.01292.x. PMID 22233397
- [Background] Hargrove JB, Bennett RM, Clauw DJ. Long-term outcomes in fibromyalgia patients treated with noninvasive cortical electrostimulation. Arch Phys Med Rehabil. 2012 Oct;93(10):1868-71. doi: 10.1016/j.apmr.2012.04.006. Epub 2012 Apr 21. PMID 22525670